CLINICAL TRIAL: NCT00312039
Title: A 14 Day Randomized, Double-blind, Study of Once Daily Elvucitabine Versus Lamivudine in Participants With a Documented M184V Mutation
Brief Title: Study of Once Daily Elvucitabine Versus Lamivudine in Participants With a Documented M184V Mutation
Acronym: Resistance
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACH443-014A
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: HIV Infections
Keywords: HIV-1; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — dexelvucitabine; Lamivudine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Elvucitabine
- B (Active Comparator)
  Interventions: Drug: Lamivudine

INTERVENTIONS:
Drug: Elvucitabine — Elvucitabine 10 mg QD for 14days
  Arms: A
Drug: Lamivudine — Lamivudine 300 mg QD for 14 days
  Arms: B

SUMMARY:
Human immunodeficiency virus (HIV)-1 infected participants receiving long-term therapy with lamivudine or emtricitabine (nucleoside reverse transcriptase inhibitors [NRTIs]) are at risk for the development of a mutation at position M184 on the HIV reverse transcriptase gene. This mutation confers resistance to both drugs (>100 fold increase in the concentration of drug producing 50% inhibition [IC50]).

In-vitro studies with elvucitabine have shown that HIV-1 isolates with the M184V mutation show only a 10-fold increase in IC50 as compared to wild type HIV-1. Alexion Pharmaceuticals Inc. intention is to demonstrate that 10 milligrams (mg) of elvucitabine, administered once per day for 14 days with continued background anti-HIV-1 medications, will demonstrate a fall in HIV-1 ribonucleic acid (RNA) plasma levels, as compared to baseline. The data from this study will guide dosing in future long-term studies in HIV-1 infected participants with the M184V mutation.

DETAILED DESCRIPTION:
This was a Phase 2a, 14-Day randomized, double-blind, comparative viral kinetic study of10 mg elvucitabine as compared to lamivudine that was administered once daily (QD) to HIV-1 infected participants with a documented M184V variant. This study also demonstrated the antiviral activity as well as the assessment of safety of the elvucitabine therapy

Participants must be receiving a stable antiretroviral regimen (defined as no change in antiretroviral therapy for at least 4 weeks prior to randomization) that includes lamivudine or emtricitabine. At 72 hours prior to randomization, only lamivudine or emtricitabine will be stopped for washout; participants will continue to receive the other drugs in their prescribed regimen (background antiretroviral therapy) during the 72-hour washout period. Participants will then be randomized to receive blinded elvucitabine or lamivudine in a 1:1 ratio and continue to receive their prescribed background antiretroviral therapy for 14 days on an outpatient basis. Participants will be followed for an additional 14 days post-treatment for safety unless they enroll in the ACH443-018 extension study where they will continue to be treated and followed for safety.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable HIV-1 infected participants
* Ages >18 and <65 years
* Documented M184V mutation
* CD4 cell count >100 cells/mL
* Plasma HIV-1 RNA levels >5000 and <150,000 copies/milliliter (mL)
* Currently receiving lamivudine or emtricitabine
* Other hematologic and metabolic parameters must be met.
* Provide written informed consent
* Other inclusion criteria apply.

Exclusion Criteria:

* Hepatitis B antigen positive
* HIV-1 genotype positive for more than or equal to 4 protease mutations
* HIV-1 genotype positive for more than or equal to 2 non-nucleoside reverse transcriptase inhibitor (NNRTI) mutations
* Previous therapy with cytotoxic or myelosuppressive drugs in the past 3 months
* Evidence or history of cirrhosis
* Women who are pregnant or breast feeding
* Other exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-03-31 (Actual); Primary Completion 2007-10-31 (Actual); Study Completion 2007-10-31 (Actual)

PRIMARY OUTCOMES:
Reduction In Viral Load | 14 days

SECONDARY OUTCOMES:
Number of Participants with a Treatment Adverse Event | 14 days

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Clinical Trial Site, Birmingham, Alabama
  - Clinical Trial Site, Sacramento, California
  - Clinical Trial Site, Miami, Florida
  - Clinical Trial Site, Orlando, Florida
  - Clinical Trial Site, West Palm Beach, Florida
  - Clinical Trial Site, Atlanta, Georgia
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Cincinnati, Ohio